CLINICAL TRIAL: NCT02623608
Title: Acute Metabolic Challenge for the Assessment of Cardiometabolic Protective Effects of Foods
Brief Title: Effects of Functional Ingredients in an Acute Metabolic Challenge Context
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Vinnova (Other Government); Antidiabetic Food Centre AFC (Unknown)
Responsible Party: Principal Investigator, Juscelino Tovar, Project Leader, Lund University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: AFC-JT-Ac.Ch
Record Dates: First submitted 2015-12-03; First posted 2015-12-07 (Estimated); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Metabolic Syndrome
Keywords: type 2 diabetes risk; cardiovascular disease risk
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- High fat meal (Experimental): Subjects eat a high fat breakfast (reference breakfast) at 7:30 am. The meal contains 50 g fat and 900 kcal. Blood samples are taken before the breakfast and every 30 min postprandial for 4 h.
  Interventions: Other: Reference breakfast
- High fat meal + Active Ingredient 1 (Experimental): Subjects eat the same high fat breakfast with the "active ingredient 1" at 7:30 am. The meal contains 50 g fat and 900 kcal. Blood samples are taken before the breakfast and every 30 min postprandial for 4 h.
  Interventions: Other: Active Ingredient 1
- High fat meal + Active Ingredient 2 (Experimental): Subjects eat the same high fat breakfast with the "active ingredient 2" at 7:30 am. The meal contains 50 g fat and 900 kcal. Blood samples are taken before the breakfast and every 30 min postprandial for 4 h.
  Interventions: Other: Active Ingredient 2
- High fat meal + Active Ingredient 3 (Experimental): Subjects eat the same high fat breakfast with the "active ingredient 3" at 7:30 am. The meal contains 50 g fat and 900 kcal. Blood samples are taken before the breakfast and every 30 min postprandial for 4 h.
  Interventions: Other: Active Ingredient 3
- High fat meal + Active Ingredient 4 (Experimental): Subjects eat the same high fat breakfast with the "active ingredient 4" at 7:30 am. The meal contains 50 g fat and 900 kcal. Blood samples are taken before the breakfast and every 30 min postprandial for 4 h.
  Interventions: Other: Active Ingredient 4

INTERVENTIONS:
Other: Reference breakfast — A high fat, high calorie breakfast
  Arms: High fat meal
Other: Active Ingredient 1 — A high fat, high calorie breakfast including the Active Ingredient 1
  Arms: High fat meal + Active Ingredient 1
Other: Active Ingredient 2 — A high fat, high calorie breakfast including the Active Ingredient 2
  Arms: High fat meal + Active Ingredient 2
Other: Active Ingredient 3 — A high fat, high calorie breakfast including the Active Ingredient 3
  Arms: High fat meal + Active Ingredient 3
Other: Active Ingredient 4 — A high fat, high calorie breakfast including the Active Ingredient 4
  Arms: High fat meal + Active Ingredient 4

SUMMARY:
After an energy-rich meal the blood levels of glucose and lipids undergo a marked temporary increase, triggering a wave of oxidative stress due to the appearance of excess free radicals in adipose and muscle tissues. Elevated postprandial hypertriglyceridemia has been associated with increased risk of cardiovascular disease and type 2 diabetes. Hence, postprandial changes in different circulating biomarkers are potential predictors of cardiometabolic risk. In addition to the possibility of evaluating acute variations in metabolic risk markers in response to different types of fat, the metabolic challenge approach may serve as a challenge-meal background in order to reveal possible beneficial effects of specific food ingredients. In this study, circulating cardiometabolic disease-related biomarkers, including endotoxemia, will be assessed postprandially in search for beneficial actions of particular functional food ingredients consumed in combination with a high-fat meal.

DETAILED DESCRIPTION:
The study will be carried out in a group of healthy mature subjects with overweight and normal fasting blood glucose values.

A randomized crossover design will be followed, in which the postprandial metabolic responses to a high fat breakfast (HF) will be compared with those registered after an identical breakfast containing a functional ("active") ingredient. Each meal will be tested in an independent experimental session. Experimental sessions will take place with1 week interval. The study will be carried out at the Food for Health Laboratory, Food for Health Science Centre - Lund University (Medicon Village, Lund).

The volunteers will consume the challenge HF alone and with 4 active ingredients, i.e. each volunteer will undergo five experimental sessions. Additionally, the plan contemplates an initial information visit that includes the screening of fasting blood glucose. In total, each volunteer completing the study will pay six visits to the Food for Health Laboratory.

Based on the results from the above-described phase, a second step of the study will focus on the impact of the order of consumption -i.e. "active ingredient" before HF and vice versa on cardiometabolic risk outcomes, as a way to optimize putative protective actions.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI between 25 and 30)
* fasting blood glucose value ≤ 6.1 mmol/l.

Exclusion Criteria:

* treatment for dyslipidemia
* treatment for hypertension

Ages: 50 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of postprandial triglyceridemia (0-4h) after each intervention, compared to the reference meal | 4 hours postprandial
  plasma triglycerides are measured pre-meal and at various post-meal intervals for up to for 4 hours. The area under curve (AUC) is calculated and compared to AUC following the reference meal.

SECONDARY OUTCOMES:
AUC of postprandial endotoxemia, i.e. lipopolysaccharide (LPS) concentrations (0-4h) after each intervention, compared to the reference meal | 4 h postprandial
  plasma LPS is measured pre-meal and and at various post-meal intervals for up to for 4 hours. AUC is calculated and compared to AUC recorded for the reference meal.
Area under the curve of postprandial glycemia (0-4h) after each intervention, compared to the reference meal | 4 hours postprandial
  plasma glucose is measured pre-meal and and at various post-meal intervals for up to for 4 hours. AUC is calculated and compared to AUC recorded after the reference meal.

CONTACTS AND LOCATIONS:
Overall Officials: Juscelino Tovar, PhD, Study Director — Lund University
Locations (1):
- Food for Health Science Centre. Lund University Medicon Village, Lund, Sweden

REFERENCES:
- [Background] O'Keefe JH, Bell DS. Postprandial hyperglycemia/hyperlipidemia (postprandial dysmetabolism) is a cardiovascular risk factor. Am J Cardiol. 2007 Sep 1;100(5):899-904. doi: 10.1016/j.amjcard.2007.03.107. Epub 2007 Jun 26. PMID 17719342
- [Background] Johnston KL, Clifford MN, Morgan LM. Coffee acutely modifies gastrointestinal hormone secretion and glucose tolerance in humans: glycemic effects of chlorogenic acid and caffeine. Am J Clin Nutr. 2003 Oct;78(4):728-33. doi: 10.1093/ajcn/78.4.728. PMID 14522730
- [Background] Strassburg K, Esser D, Vreeken RJ, Hankemeier T, Muller M, van Duynhoven J, van Golde J, van Dijk SJ, Afman LA, Jacobs DM. Postprandial fatty acid specific changes in circulating oxylipins in lean and obese men after high-fat challenge tests. Mol Nutr Food Res. 2014 Mar;58(3):591-600. doi: 10.1002/mnfr.201300321. Epub 2013 Oct 14. PMID 24127338
- [Background] Herieka M, Erridge C. High-fat meal induced postprandial inflammation. Mol Nutr Food Res. 2014 Jan;58(1):136-46. doi: 10.1002/mnfr.201300104. Epub 2013 Jul 12. PMID 23847095
- See also: Food for Health Science Centre/Antidiabetic Food Centre, hosts of the study — https://portal.research.lu.se/portal/en/projects/antidiabetic-food-centre(3a9bae87-b64a-49f5-97a4-868a8bb776ae).html
- See also: Published results — https://doi.org/10.1016/j.jff.2017.09.019
- See also: Published results — https://doi.org/10.1016/j.jff.2019.103443